CLINICAL TRIAL: NCT05400096
Title: Body Image, Psychological Distress, Shame and Disordered Eating in Patients in a Tier 3 Weight Management Service Receiving an Online Delivered, Group Based Compassion Focused Therapy (CFT) Informed Psychological Intervention
Brief Title: Psychological Wellbeing in Clients in Tier 3 Weight Management Service
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DClinPsych2020UTartilaite
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Psychological Distress; Obesity; Disordered Eating; Shame; Body Image
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CFT based online group intervention (Experimental): The group will consist of 12 weekly 1.15h long online sessions.
  Interventions: Other: Psychological therapy

INTERVENTIONS:
Other: Psychological therapy — The protocol for the group will be developed collaboratively between the chief researcher and the supervisor based in the weight management service. The protocol will contain Compassion Focused Therapy (CFT) based therapeutic approaches, but the group will integrate some Acceptance and Commitment Therapy (ACT) concepts.

SUMMARY:
This study aims to conduct an initial, single case investigation of changes in feelings of shame, overall psychological wellbeing, body image and disordered eating in patients in naturalistic setting, Tier 3 weight management service, following CFT based, online group intervention that runs for 12 weeks.

DETAILED DESCRIPTION:
Tier 3 weight management services are led by multidisciplinary teams (MDTS) what usually include physicians, dieticians, nurses, physiotherapist, psychiatrists, and psychologists. In the service where the study is conducted referrals to psychology are often made by a dietician. The psychologist in the service also accepts self referrals from patients either during initial assessment with dieticians or at any point of their journey in the service. The psychology pathway is "opt-in", in other words, only patient who actively express interest, motivation and wish to make use of the additional psych resource and accepted.

The participants will be offered the intervention by the group facilitating clinician (who is a part of care team). Initially the principal supervisor was meant to facilitate group intervention, but because the principal supervisor is going on maternity leave the group will be facilitated by a qualified substitute clinician. This clinician will offer an assessment of needs to all patients referred for psychological support. The clinician will act as a gatekeeper and will offer CFT based group intervention when clinically and ethically appropriate (see the exclusion and inclusion criteria below). Taking part in the intervention and signing up for the research will not affect the care patients receive from MDT in the service.

ELIGIBILITY:
Inclusion Criteria:

* adults with BMI over 30 who have been referred to Tier 3 weight management service.
* Adults with BMI over 25 with Diabetes who have been referred to Tier 3 weight management service.

Exclusion Criteria:

* group intervention not considered clinically appropriate, following specialist assessment of needs
* not being able to commit to 12-week intervention
* severe interpersonal difficulties that would be disruptive to other group's participants
* moderate to severe learning difficulties
* current alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Experiential Shame Scale | 20 weeks
  25 items questionnaire. Rated on 4 point Likert scale from 1 (not at all) to 4 (very much).Higher scores indicate higher shame. Minimum of total scores-25, Maximum of total scores- 100.
Clinical Outcomes in Routine Evaluation 10 | 20 weeks
  10 items questionnaire. Items on the CORE measures are scored from zero to four, with higher scores indicating greater levels of distress. Scores of the CORE-10 can be divided into categories of distress: Healthy (0-5), low (6-10), mild (11-14), moderate (15-19), moderate-to-severe (20-24), and severe (25 and above). The maximum of total scores-40, the minimum of total score-0.
Disordered Eating Questionnaire | 20 weeks
  In part A answers are given on a 5-point frequency scale, the alternatives being never, 1-2 per week, 3-4 per week, every day, more than once a day. In part B the answers are given on a 7-point likert scale ranging from 1 (not at all) to 7 (absolutely). Section A consists of 18 items which evaluate the frequency with which the subject adopts a series of disordered eating behaviors. Section B has 6 items dealing with worries and intrusive thoughts regarding weight, food, calories, physical fitness. The unifactorial structure includes all the items from section A, with the exception of the 4 items concerning purging behaviours and all the items from section B. Adding up the scores of all the items included in the factor, a scale score is obtained whose reliability (measured using Cronbach's alpha) is equal to 0.90.
  The frequency of purging behaviours is calculated separately by adding the frequencies given in the relative 4 items not included in the scale score.
The Three-Factor Eating Questionnaire-Revised | 20 weeks
  The instrument has 18 items. The responses are given in likert like scale where points range from 1-4, the final question asks to self rate from 1-8. The maximum of total possible (raw) scores is 76, the minimum is 18. The instrument consists of 3 scales: Cognitive Restraint, Uncontrolled Eating and Emotional Eating Scale. Higher scores in the respective scales are indicative of greater cognitive restraint, uncontrolled, or emotional eating. The raw scale scores are standardized to a 0-100 scale using a formula.
The Body Appreciation Scale-2 | 20 weeks
  10-item scale. The items are rated along a 5-point scale (1 = never, 2 = seldom,3= sometimes,4= often,5= always) and are averaged to obtain an overall body appreciation score. Higher scores reflect greater body appreciation. The maximum of total possible scores is 50, the minimum is 10.

OTHER OUTCOMES:
Experience of the intervention after it has ended | 20 weeks
  1. What would you say had the biggest impact on you as the result of the work you did in the group?
  2. How did the work during the group affect your relationship with your body if at all?
  3. How did the work during the group affect your relationship with food if at all?
  4. Has anything else happened in your life in the last 12 weeks that had an impact on your psychological wellbeing, sense of shame, relationship with food or your body?
  5. Is there anything else about your experience of the work you did in the group that is important and that you would like to mention?

IPD SHARING:
Plan to Share IPD: No